CLINICAL TRIAL: NCT04693988
Title: Early Case Management on Recovery From a Cardiac Event in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Sherrie Khadanga, Assistant Professor of Medicine, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001090; P20GM103644 (NIH)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Rehabilitation
Keywords: Secondary Prevention, Women's cardiovascular disease, case management
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case management (Experimental): Patient receives case management while in hospital.
  Interventions: Behavioral: Case Management
- Usual Care (No Intervention): This control condition does not receive intervention of case management

INTERVENTIONS:
Behavioral: Case Management — a case manager is available by phone to assist patient with attending cardiac rehabilitation sessions as well as provide advice about cardiac symptoms and behavioral life style changes
  Arms: Case management

SUMMARY:
Outpatient cardiac rehabilitation (CR) is an exercise-based lifestyle program for patients who have experienced a myocardial infarction, systolic heart failure, percutaneous revascularization or cardiac surgery. CR plays a key role in secondary prevention, which is the prevention of subsequent cardiac events. CR has been shown to reduce both cardiovascular mortality and one year hospital readmissions as well as improve quality of life, exercise capacity, and physical function. Although the benefits have been clearly established for cardiac patients, women are much less likely to attend CR than men. Based upon our own preliminary data (and the medical literature), attendance at CR is determined by factors that vary in their importance between men and women. These findings demonstrate that older age and poor social support are particular barriers to CR participation in women. This information can guide efforts to increase CR participation and adherence in women, areas which have received little study.

Case management (CM) has been effective at reducing cardiovascular risk and reducing hospitalizations amongst cardiac patients. Further, CM has been effective at promoting attendance in a variety of health related programs (for example, diabetes treatment or cocaine dependence treatment). The primary aim in this randomized controlled trial is to examine the efficacy of early CM to promote participation and adherence in CR. The CM model can identify individualized determinants of health and social needs to identify potential barriers which may hinder CR enrollment. Additionally, the case manager will conduct a home visit and provide individual counseling to address lifestyle changes including physical activity. Thus, a component of CR and physical activity can be still be delivered for those unable to attend CR. The concept of CM to improve CR participation and adherence has not been specifically tested in women, a vulnerable patient population. This intervention, therefore, has the potential to increase utilization of CR and significantly improve health outcomes in female cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

1. A cardiac rehabilitation qualifying condition including: A recent myocardial infarction or coronary revascularization or heart valve replacement or repair, stable angina, or congestive heart failure (ejection fraction <35%)
2. Lives in and plans to remain in the greater Burlington, Vermont area for the next year.

Exclusion Criteria:

1. Severe dementia
2. Advanced cancer, advanced frailty, or other longevity-limiting systemic disease
3. Severe life threatening ventricular arrhythmias unless adequately controlled (e.g. intracardiac defibrillator)
4. Exercise-limiting non-cardiac disease such as severe arthritis, past stroke leading to paralysis
5. Participation in cardiac rehab within the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Rehabilitation Participation | within 4 months of the intake assessment
  Attendance of at least 1 session
Cardiac Rehabilitation Adherence | within 4 months of the intake assessment
  Number of cardiac rehabilitation sessions completed out of a possible 36

SECONDARY OUTCOMES:
Changes in Physical Activity | within 4 months of the intake assessment
  Changes in fitness level (step count) will be measured from intake to completion of the intervention (4 months after intake)
Changes in Quality of Life | within 4 months of the intake assessment
  Changes in perceived quality of life (MacNew) questionnaires will be measured from intake to completion of the intervention (4 months after intake)
Changes in Self Reported Physical Function | within 4 months of the intake assessment
  Changes in perceived physical function (Medical Outcomes Study Short Form-36) will be measured from intake to completion of the intervention (4 months after intake)
Changes in Depression | within 4 months of the intake assessment
  Changes in depression (Patient Health Questionnaire-9) will be measured from intake to completion of the intervention (4 months after intake)
Changes in Anxiety | within 4 months of the intake assessment
  Changes in anxiety (Generalized Anxiety Disorder questionnaire) will be measured from intake to completion of the intervention (4 months after intake)

OTHER OUTCOMES:
Maintenance of Physical Activity following Intervention | From completion of intervention (4 months) to follow up (one year)
  Changes in step count will be measure from intervention completion until follow-up (8 months after intervention completion)
Maintenance of Quality of Life following Intervention | From completion of intervention (4 months) to follow up (one year)
  Changes in perceived quality of life (MacNew questionnaire) will be measured from intervention completion until follow-up (8 months after intervention completion)
Maintenance of Self Reported Physical Function following Intervention | From completion of intervention (4 months) to follow up (one year)
  Changes in perceived physical function (Medical Outcomes Study Short Form-36) will be measured from intervention completion until follow-up (8 months after intervention completion)
Maintenance of Depression following Intervention | From completion of intervention (4 months) to follow up (one year)
  Changes in mental health (Patient Health Questionnaire-9) will be measured from intervention completion until follow-up (8 months after intervention completion)
Maintenance of Anxiety following Intervention | From completion of intervention (4 months) to follow up (one year)
  Changes in mental health (Generalized Anxiety Disorder questionnaire) will be measured from intervention completion until follow-up (8 months after intervention completion)
Health Care Contacts | One year period starting at intake assessment
  Combined measure of number of Emergency Department visits and overnight hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No